CLINICAL TRIAL: NCT07352488
Title: Effect of Modified Shenling Baizhu Powder on Allergic Asthma With Spleen Deficiency and Dampness Accumulation Syndrome: A Multicenter, Randomized Controlled Trial
Brief Title: Modified Shenling Baizhu Powder for Allergic Asthma With Spleen Deficiency and Dampness Accumulation Syndrome
Acronym: mSLBZP-Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024YFC3505302
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Allergic Asthma
Keywords: Allergic asthma; Modified Shenling Baizhu Powder; Spleen Deficiency and Dampness Accumulation Syndrome; Randomized controlled trial
MeSH Terms: interventions — Budesonide; Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive Modified Shenling Baizhu Powder in addition to Budesonide and Formoterol Fumarate Powder for Inhalation.
  Interventions: Drug: Modified Shenling Baizhu Powder; Drug: Budesonide and Formoterol Fumarate Powder for Inhalation
- Control group (Placebo Comparator): The control group will receive a placebo in addition to Budesonide and Formoterol Fumarate Powder for Inhalation.
  Interventions: Drug: Placebo; Drug: Budesonide and Formoterol Fumarate Powder for Inhalation

INTERVENTIONS:
Drug: Modified Shenling Baizhu Powder — Modified Shenling Baizhu Powder will be taken twice daily.
  Arms: Experimental group
Drug: Placebo — The placebo will be taken twice daily.
  Arms: Control group
Drug: Budesonide and Formoterol Fumarate Powder for Inhalation — Budesonide and Formoterol Fumarate Powder for Inhalation will be taken twice daily.

SUMMARY:
Allergic asthma is a common allergic disease characterized by a protracted disease course and recurrent episodes, which severely impairs patients' physical and mental health. There is a paucity of high-quality clinical evidence in the treatment of allergic asthma with traditional Chinese medicine (TCM). This study will enroll patients who are persistent allergic asthma with spleen deficiency and dampness accumulation syndrome. A multicenter, randomized, double-blind, placebo-controlled trial design is adopted. The experimental group will receive Modified Shenling Baizhu Powder in addition to Budesonide and Formoterol Fumarate Powder for Inhalation, while the control group will receive a placebo in addition to the same inhalation therapy. Both groups will undergo an 8 week of treatment followed by a 12 week of follow-up. The primary outcome is Asthma Control Test scores, and the secondary outcomes include acute exacerbations, Asthma Control Questionnaire scores, Asthma Quality of Life Questionnaire scores, pulmonary function, airway inflammatory markers, clinical symptom scores, serum inflammatory markers, immune markers, and use of controller medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are persistent allergic asthma.
* Patients who meet the diagnostic criteria for the spleen deficiency and dampness accumulation syndrome.
* Patients who are aged between 18 and 80 years.
* Patients who voluntarily accept the treatment and sign the informed consent form.

Exclusion Criteria:

* Patients who have chronic obstructive pulmonary disease, interstitial lung disease, bronchiectasis, allergic bronchopulmonary aspergillosis, eosinophilic granulomatosis with polyangiitis , active pulmonary tuberculosis, or pulmonary embolism, etc.
* Patients who have severe cardiovascular or cerebrovascular diseases.
* Patients who have severe liver or kidney diseases.
* Patients who have a history of tumor.
* Patients who have cognitive impairment or psychiatric disorders.
* Patients who are pregnant or breastfeeding.
* Patients who are allergic to medication(s) used.
* Patients who participated in another clinical trial within one month prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test scores | At baseline, week 4 and week 8 of treatment, and week 12 of follow-up.
  To be measured by Asthma Control Test.

SECONDARY OUTCOMES:
Acute exacerbation | At baseline, week 4 and week 8 of treatment, and week 12 of follow-up.
  To be measured by the frequency and severity of acute exacerbation, and the time to first acute exacerbation.
Asthma Control Questionnaire scores | At baseline, week 4 and week 8 of treatment, and week 12 of follow-up.
  To be measured by Asthma Control Questionnaire.
Asthma Quality of Life Questionnaire scores | At baseline, week 4 and week 8 of treatment, and week 12 of follow-up.
  To be measured by Asthma Quality of Life Questionnaire.
Pulmonary function | At baseline, week 8 of treatment, and week 12 of follow-up.
  To be measured by pulmonary function test.
Airway inflammatory markers | At baseline, week 8 of treatment, and week 12 of follow-up.
  To be measured by fractional exhaled nitric oxide.
Clinical symptom scores | At baseline, week 4 and week 8 of treatment, and week 12 of follow-up.
  To be measured by clinical symptom questionnaire.
Serum inflammatory markers | At baseline, week 4 and week 8 of treatment.
  To be measured by blood eosinophil count, total serum IgE, IL-4, IL-5, TNF-α, etc.
Immune markers | At baseline, week 4 or week 8 of treatment.
  To be measured by CD4+, CD8+, CD4+/CD8+, Th17, and Treg.
Use of controller medications | At baseline, week 4 and week 8 of treatment, and week 12 of follow-up.
  To be measured by the usage of bronchodilator and glucocorticoid.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No